CLINICAL TRIAL: NCT02058498
Title: Increasing Physical Activity in Post Liver Transplant Patients
Brief Title: Increasing Activity in Liver Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jennifer L. Serotta, A.R.N.P., ARNP, FNP-BC, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13-004699
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Liver Transplant
Keywords: Liver transplant; Physical Activity; Quality of Life
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liver Transplant Patients (Experimental): Participants will be provided physical activity walking instructions and asked to record their daily activity on an activity log.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Participants will be provided physical activity walking instructions and asked to record their daily activity on an activity log. Participants will be given the International Physical Activity Questionnaire and asked about their quality of life at baseline, at 6 weeks and at 4 months.

SUMMARY:
Will adult liver transplant patients who are provided with physical activity (walking) instructions increase their physical activity and perceive an improved quality of life?

ELIGIBILITY:
Inclusion criteria:

* Adult patients 18-65 years of age who receive a liver transplant at Mayo Clinic Jacksonville.
* Adult patients who are 5-21 days post liver transplant.
* Must be followed by Mayo Clinic Jacksonville at 4 months postoperatively.
* Approved by a hepatologist and/or transplant surgeon to participate.

Exclusion criteria:

* Patients with active infections
* Patients with encephalopathy or cognitive dysfunction
* Patients who receive a combined liver-kidney transplant
* Patients with severe debility
* Patients who require assistance to ambulate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Serotta, ARNP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Mayo Clinic in Jacksonville, Florida. Data were collected from April 2014 to September 2014.
Period: Overall Study
Arm/Group | Liver Transplant Patients
Started | 12
6 Weeks | 8
Completed | 8
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Liver Transplant Patients
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Measured by the International Physical Activity Questionnaire (IPAQ)
Description: The IPAQ calculates the metabolic equivalent (MET) score by asking participants the days and minutes exercised in three categories of intensity (vigorous, moderate, and walking) during the previous one week. The following formula is used to calculate the MET: MET=8(vigorous activity) (minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes).
Time Frame: Baseline, 6 weeks
Measure: Median (Full Range); unit: MET
Arm/Group | Liver Transplant Patients
Number analyzed (Participants) | 8
MET
  Baseline | 407 [99 to 14,826]
  6 weeks | 1711 [462 to 2479]

2. Secondary Outcome: Quality of Life at Baseline, 6 Weeks, and 4 Months
Description: Participants reported their perceived quality of life using a scale 1 - 10, with 1 being the worst and 10 being the best.
Time Frame: Baseline, 6 weeks, 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liver Transplant Patients
Number analyzed (Participants) | 8
units on a scale
  Baseline | 5.5 (2.5)
  6 Weeks | 8.25 (1.6)
  4 months | 8.3 (1.6)
Statistical Analysis 1: Comparison: Liver Transplant Patients; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Patients Who Document Their Physical Activity
Description: 8 participants documented their physical activity at 6 weeks. 6 participants documented their physical activity at 4 months.
Time Frame: Baseline to 6 weeks, repeated measure at 4 months
Measure: Number; unit: participants
Arm/Group | Liver Transplant Patients
Number analyzed (Participants) | 8
participants
  6 weeks | 8
  4 months | 6

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Liver Transplant Patients
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes